CLINICAL TRIAL: NCT04363463
Title: Impact of Prone Position in Patients Under Spontaneous Breathing on Intubation or Non-invasive Ventilation or Death Incidence During COVID-19 Acute Respiratory Distress
Acronym: PROVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHRO-2020-09
Record Dates: First submitted 2020-04-22; First posted 2020-04-27 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: COVID19; Oxygen Therapy; Prone Position; Spontaneous Ventilation; Respiratory Distress Syndrome
Keywords: COVID19; Oxygen therapy; Prone position; Spontaneous ventilation; Acute respiratory failure
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: Randomized controlled multicenter trial Ratio 1:1
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional positioning (No Intervention): semi-seated in bed or seated in a chair during the day. The prone position is not allowed during the day (it is allowed at night if it is the natural sleeping position).
- Interventional positioning : prone position (Experimental): Two sessions minimum of prone position over the day. With a total objective of at least 2h30 of cumulated duration over the day. The objective is to spend as much time as possible in prone position if the patient tolerates it well.
  Interventions: Other: prone position

INTERVENTIONS:
Other: prone position — Two sessions minimum of prone position over the day. With a total objective of at least 2h30 of cumulated duration over the day. The objective is to spend as much time as possible in prone position if the patient tolerates it well.
  Arms: Interventional positioning : prone position

SUMMARY:
The SARS-Cov2 viral pandemic is responsible for a new infectious disease called COVID-19 (CoronaVIrus Disease), is a major health problem. Respiratory complications occur in 15 to 40%, the most serious is acute respiratory distress syndrome (ARDS).

The management of COVID-19 is essentially symptomatic with respiratory oxygen supplementation in mild forms to invasive mechanical ventilation in the most severe forms.

Prone position (PP) reduced mortality in patients with ARDS in intensive care. Ding et al showed that PP and high flow oxygenation reduced the intubation in patients with moderate to severe ARDS.

The investigators hypothesize that the use of PP in spontaneously ventilation patients under oxygen standard could decrease incidence of intubation or non-invasive ventilation or death compared to conventional positioning management in medical departments.

DETAILED DESCRIPTION:
This is a multicenter randomized controlled study. 400 patients with COVID-19 documentation and undergoing oxygen therapy will be randomly assigned, with a 1:1 ratio, to conventional positioning or repeated prone sessions.

The control group will have conventional positioning: semi-seated in bed or seated in a chair. The prone position is not allowed during the day (it is allowed at night if it is the natural sleeping position).

The intervention group will have:

* Two sessions minimum of prone position over the day. With a total objective of at least 2h30 of cumulated duration over the day. The objective is to spend as much time as possible in prone position if the patient tolerates it well.
* The maximum of prone position at night. Patients must be able to take position by themselves or with minimal assistance. The rails will be positioned in order to prevent falling out of bed. The patient will be free to choose his preferred prone position as long as the back is not compressed

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 85 years old
* With COVID-19 documentation
* Undergoing oxygen therapy (nasal cannula, medium or high concentration mask or high flow nasal oxygen therapy)
* Able to move to PP by him/herself or with minimal assistance
* Written consent
* Hospitalized in COVID medical department for less than 72 hours

Exclusion Criteria:

* Pregnant (positive pregnancy test during screening) or breastfeeding women
* Patient on long-term oxygen therapy or Continuous Positive Airway Pressure (CPAP) or Non-Invasive Ventilation (NIV) at home
* Chronic Obstructive Pulmonary Disease (COPD) Patient stage 3 or 4
* Patient with known chronic diffuse interstitial lung disease
* Patient with neuromuscular pathology
* Contraindication to the PP (recent thoracic trauma, pneumothorax, orthopaedic fracture preventing mobilization, ...)
* Deep vein thrombosis of the lower limbs or pulmonary embolism with effective anticoagulation for less than 48 hours
* Hemodynamic instability (MAP < 65 mm Hg) persisting for more than 1 hour
* Respiratory rate greater than 40 cycles per minute
* Excessive use of accessory respiratory muscles (as judged by the clinician)
* Indication for curative NIV (acute pulmonary edema or acute hypercapnic respiratory failure)
* Intestinal Occlusive Syndrome
* Patient unable to protect upper airway
* Inability to understand French or to follow instructions for the prone position.
* Person under guardianship
* Protected Majors
* Not affiliated to French social security
* Decision not to forgo life sustaining therapy
* Patient discharged from an intensive care unit and has been treated by invasive or non-invasive mechanical ventilation at 2 pressure levels during the resuscitation stay.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Percent age of patients who will have endotracheal intubation or non-invasive ventilation at two pressure levels and/or die, in each of the 2 randomization groups. | Day 28
  To show that PP in spontaneously ventilation patients could reduce the risk of acquiring the following event (composite endpoint):
  * Endotracheal intubation
  * Or non-invasive ventilation (NIV) with two pressure levels
  * And/or death

SECONDARY OUTCOMES:
Duration in days for the change of 2 points on the WHO ordinal scale | Day 28
  Show that the use of prone position improves the WHO ordinal scale score by 2 points faster (after randomization)
Rate (%) of intubation and invasive ventilation in the 2 randomization groups. | Day 28
  Show that prone position with spontaneous ventilation reduces the need for endotracheal intubation and invasive mechanical ventilation
Rate (%) of non-invasive ventilation at two pressure levels in the 2 randomization groups | Day 28
  Show that prone position with spontaneous ventilation reduces the use of non-invasive ventilation at two pressure levels
Duration of oxygen therapy in the 2 randomization groups. | Day 28
  Show that prone position in spontaneous ventilation reduces the time under oxygen therapy.
Duration of hospitalization in the 2 randomization groups. | Day 28
  Show that prone position reduces the length of hospitalization.
Hospital mortality and mortality at D28 in the 2 randomization groups | Day 28
  Compare the hospital mortality of the 2 groups
Rate (%) of need for transfer to intensive care unit | Day 28
  Compare the incidence of the need for resuscitation transfer between the two groups.
Rate (%) of use of non-invasive ventilation at two pressure levels, intubation throughout the entire stay when the stay is longer than 28 days. | 1 year
  Compare the impact of the use of non-invasive ventilation and intubation on the entire hospital stay when the hospital stay is longer than 28 days between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Anh NAY, Dr, Study Chair — CHR Orléans
Locations (19):
- France (18):
  - CH de Blois, Blois
  - CH de DAX, Dax
  - CHD de VENDEE, La Roche-sur-Yon
  - CH de LA ROCHELLE, La Rochelle
  - CH Le Mans, Le Mans
  - CH Mont de MArsan, Mont-de-Marsan
  - CHR d'Orléans - Service Pneumologie, Orléans
  - CHR d'Orleans - Service Maladies Infectieuses, Orléans
  - HOPITAL LARIBOISIERE - Service diabétologie, endocrinologie, nutrition, Paris
  - Hopital Européen Georges Pompidou, Paris
  - Hopital Lariboisiere - Medecine Interne, Paris
  - Hopital Lariboisiere, Paris
  - CH de PERPIGNAN - Service Maladies infectieuses, Perpignan
  - Centre Hospitalier Intercommunal de Cornouaille - Quimper Concarneau, Quimper
  - CHRU de Tours - Service Médecine interne et immunologie Clinique, Tours
  - CHRU de Tours - Service Pneumologie, Tours
  - CHRU DE TOURS - Service Médecine interne et maladies infectieuses, Tours
  - CH Bretagne Atlantique, Vannes
- centre Hospitalier Princesse Grace, Monaco, Monaco

REFERENCES:
- [Background] Murthy S, Gomersall CD, Fowler RA. Care for Critically Ill Patients With COVID-19. JAMA. 2020 Apr 21;323(15):1499-1500. doi: 10.1001/jama.2020.3633. No abstract available. PMID 32159735
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Derived] Nay MA, Hindre R, Perrin C, Clement J, Plantier L, Seve A, Druelle S, Morrier M, Laine JB, Colombain L, Corvaisier G, Bizien N, Pouget-Abadie X, Bigot A, Jamard S, Nyamankolly E, Planquette B, Fossat G, Boulain T. Prone position versus usual care in hypoxemic COVID-19 patients in medical wards: a randomised controlled trial. Crit Care. 2023 Jun 17;27(1):240. doi: 10.1186/s13054-023-04529-z. PMID 37330512
- [Derived] Nay MA, Planquette B, Perrin C, Clement J, Plantier L, Seve A, Druelle S, Morrier M, Laine JB, Colombain L, Corvaisier G, Bizien N, Pouget-Abadie X, Bigot A, Bernard L, Nyamankolly E, Fossat G, Boulain T. Does awake prone positioning prevent the use of mechanical respiratory support or death in COVID-19 patients on standard oxygen therapy hospitalised in general wards? A multicentre randomised controlled trial: the PROVID-19 protocol. BMJ Open. 2022 Jul 8;12(7):e060320. doi: 10.1136/bmjopen-2021-060320. PMID 35803621